CLINICAL TRIAL: NCT06918015
Title: A Prospective, Single-arm, Phase II Study of Zanubrutinib in Combination With GCVP (Obinutuzumab, Cyclophosphamide, Vindesine, Prednisolone) in Previously Untreated Follicular Lymphoma
Brief Title: Zanubrutinib Plus GCVP (Obinutuzumab, Cyclophosphamide, Vindesine, Prednisolone) in Previously Untreated Follicular Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yang haiyan, Chief Physician, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZGCVP
Record Dates: First submitted 2025-03-20; First posted 2025-04-09 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: BTK Inhibitors; Follicular Lymphoma; Immunochemotherapy
Keywords: BTK inhibitors; follicular lymphoma; immunochemotherapy; first-line therapy
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- zanubrutinib, obinutuzumab, cyclophosphamide, vindesine, prednisolone (Experimental): Patients receive the ZGCVP regimen (zanubrutinib, obinutuzumab, cyclophosphamide, vindesine, prednisolone) for 6 cycles at the following dose:
  1. Zanubrutinib: 160mg orally twice daily;
  2. Obinutuzumab: 1000mg intravenously on days 1, 8, and 15 of cycle 1 and on day 1 of subsequent 5 cycles;
  3. Cyclophosphamide: 750m/m2 intravenously on days 1 of every cycle;
  4. Vindesine: 3 mg/m2 (maximum dose 4 mg) intravenously on days 1 of every cycle;
  5. Prednisolone: 30mg orally three times daily on day 1-5 of every cycle.
  Interventions: Drug: ZGCVP

INTERVENTIONS:
Drug: ZGCVP — Patients receive the ZGCVP regimen (zanubrutinib, obinutuzumab, cyclophosphamide, vindesine, prednisolone) for 6 cycles at the following dose:
  1. Zanubrutinib: 160mg orally twice daily;
  2. Obinutuzumab: 1000mg intravenously on days 1, 8, and 15 of cycle 1 and on day 1 of subsequent 5 cycles;
  3. Cyclophosphamide: 750m/m2 intravenously on days 1 of every cycle;
  4. Vindesine: 3 mg/m2 (maximum dose 4 mg) intravenously on days 1 of every cycle;
  5. Prednisolone: 30mg orally three times daily on day 1-5 of every cycle. Patients achieving CR at stage II underwent observation directly; those at stage III/IV receive obinutuzumab maintenance every 8 weeks for 2 years (1000mg intravenously) until disease progression or withdrawal. Patients with disease progression during treatment switch to second-line therapy.
  Other Names: ZGCOP

SUMMARY:
Previously untreated patients with follicular lymphoma are treated with the ZGCVP regimen (zanubrutinib, obinutuzumab, cyclophosphamide, vindesine, prednisolone) for 6 cycles.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multi-center, phase II clinical study aiming at evaluating the efficacy and safety of zanubrutinib with GCVP (obinutuzumab, cyclophosphamide, vindesine, prednisolone) in untreated follicular lymphoma (FL). It includes screening (14 days before the first dose), treatment, and follow-up phases.

Screening: Recruitment subjects are grade 1-3a, stage III/IV or extensive stage II (unsuitable for radiotherapy) FL patients, with measurable lesions (short axis ≥1.5cm), meeting GELF criteria or having strong treatment desire.

Treatment: Patients receive the ZGCVP regimen for 6 cycles (21-day/cycle). Imaging evaluation was conducted at the end of every 2 cycles. Enhanced Computed Tomography (CT) and ultrasound are performed after 2 cycles of the ZGCVP regimen, while interim Positron Emission Tomography (iPET) is performed after 4/6 cycles. Bone marrow examination is required for those with initial bone marrow involvement after achieving Imaging complete response. Efficacy assessment indicators include complete response rate (CR), objection response rate (ORR), duration of response (DOR), progression free survival (PFS), overall survival (OS) and disease transformation rate according to Lugano 2014 criteria. Safety assessment indicators inlude adverse events basing on CTCAE 5.0.

Follow-up: Patients achieving CR at stage II underwent observation directly; those at stage III/IV receive obinutuzumab maintenance every 8 weeks for 2 years until disease progression or withdrawal. Patients with disease progression during treatment switch to second-line therapy.

ELIGIBILITY:
Inclusion Criteria

1. Participate in the clinical study voluntarily, fully understand and be informed of the study, sign the informed consent in person, willing to follow and be able to complete all test procedures.
2. 18-80 years old (inclusive), all genders.
3. Histopathologically confirmed grade 1-3a follicular lymphoma (FL) at stage III/IV or extensive stage II disease not suitable for radiotherapy, with at least one evaluable lesion (short axis ≥ 1.5 cm), meeting treatment indications according to GELF criteria or having a strong treatment desire.
4. No prior anti-tumor therapy, such as chemotherapy, radiotherapy, immunotherapy or biotherapy (tumor vaccine, cytokine, or growth factor controlling cancer).
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-3.
6. Adequate bone marrow and organ function, no serious hematopoietic dysfunction, abnormal heart, lung, liver, kidney function and immune deficiency.

   * Blood routine: White blood cell count ≥ 3.0×109/L, Absolute neutrophil count ≥ 1.5×109/L (use of granulocyte colony stimulating factor is permitted), Hemoglobin ≥ 9.0 g/dL (pre-transfusion or use of recombinant human erythropoietin is permitted), Platelet count ≥ 75×109/L (transfusion is permitted to reach this level). If peripheral blood abnormalities are due to lymphoma infiltration of the bone marrow or spleen, enrollment may be considered at the investigator's discretion.
   * Echocardiogram: Left ventricular ejection fraction (LVEF) ≥ 50%.
   * Liver function: serum bilirubin ≤ 2.5 times the upper limit of normal value, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal value (AST is allowed if liver is involved, ALT ≤ 5 times the upper limit of normal value).
   * Renal function: creatinine clearance ≥ 60 mL/min (estimated according to the Cockcroft-Gault formula).
   * Coagulation function: INR ≤ 1.5 times the upper limit of normal value; PT and APTT ≤ 1.5 times the upper limit of normal value.
7. Life Expectancy of at least 6 months.
8. Men and women of childbearing potential must use contraception during the study and for at least 90 days after the last dose of study medication.

Exclusion Criteria

1. Central nervous system involvement secondary to lymphoma.
2. Known severe allergic reactions to humanized or murine monoclonal antibodies, or known contraindications to any drug in the regimen.
3. History of other active malignant diseases within 2 years prior to study entry, but eligibility for inclusion: a) adequately treated carcinoma in situ of the cervix; b) local basal cell carcinoma or squamous cell carcinoma of skin; c) Pre-existing malignant disease that is under control and has undergone local radical treatment (surgical or other forms).
4. History of Human Immunodeficiency Virus (HIV) infection and/or other acquired Immunodeficiency syndrome. During screening period, patients with hepatitis B virus (HBV) surface antigen or hepatitis C virus (HCV) antibody positive must further test HBV DNA (no more than 2000 iu/ml) and HCV RNA (not exceed the method detection limit). Those ruling out active HBV or HCV infection are permitted to participate in the study. Carriers of the HBV, those with stable HBV after treatment or cured of HCV are also allowed to be enrolled.
5. Any active infections, including but not limited to bacterial, fungal or viral infections, that require systemic anti-infective treatment within 14 days prior to initiation treatment.
6. Major surgery was performed within 28 days prior to initiation treatment.
7. Combined with severe or uncontrolled disease, including but not limited to congestive heart failure, uncontrolled hypertension, unstable angina, active peptic ulcer, severe hemorrhagic diseases (such as hemophilia, von willebrand disease) or spontaneous bleeding.
8. History of stroke or intracranial hemorrhage within 6 months prior to initiation treatment.
9. Continuous treatment with strong and moderate CYP3A inhibitors or CYP3A inducers is required.
10. History of severe neurological or psychiatric disorders, including but not limited to dementia or epilepsy.
11. Conditions related to drug abuse or medical, psychological and social issues that may interfere with study participation or outcome evaluation.

    Investigator Discretion: Any patient deemed unsuitable for enrollment by the investigator.
12. Patients deemed unsuitable for the study by investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
CRR | 21days after the end of treatment
  Complete response rate

SECONDARY OUTCOMES:
ORR | 21days after the end of treatment
  Objective response rate
DOR | the time from the date of initial assessment as complete response (CR) or partial response (PR) until the date of disease progression or death from any cause, whichever occurs first, assessed up to 24 months
  Duration of response
PFS | the time from the date of initial treatment until the date of disease progression or death from any cause, whichever occurs first, assessed up to 24 months
  Progression free survival
OS | the time from the date of initial treatment until the date of death from any cause, assessed up to 24 months
  Overall survival
Disease Transformation Rate | From the first day of treatment until histological confirmation of transformation, death, or end of study follow-up, whichever occurs first, assessed up to 24 months
  The probability of histologically confirmed transformation to aggressive lymphoma among enrolled follicular lymphoma patients

OTHER OUTCOMES:
AE and SAE | from the first day of treatment until 30 days after the last treatment
  Adverse event and serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Yang, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No